CLINICAL TRIAL: NCT01431833
Title: A Phase 1 Open-Label Study With Oral TR-701 FA to Assess Pharmacokinetics and Safety in Subjects With Moderate or Severe Hepatic Impairment
Brief Title: A PK and Safety Study in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 1986-001; TR701-124 (Other: TriusRX Unique ID)
Record Dates: First submitted 2011-08-05; First posted 2011-09-12 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Matched control subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate hepatic (Experimental)
  Interventions: Drug: TR-701 FA
- Severe Hepatic (Experimental)
  Interventions: Drug: TR-701 FA
- Matched control (Experimental)
  Interventions: Drug: TR-701 FA

INTERVENTIONS:
Drug: TR-701 FA — Oral single dose 200 mg

SUMMARY:
Assess the single dose PK and safety of TR701 FA in subjects with Moderate or Severe hepatic impairment versus matched control subjects with normal hepatic function.

DETAILED DESCRIPTION:
This study will assess the single-dose pharmacokinetics (PK) and safety of TR-701 free acid (FA) in subjects with Moderate or Severe hepatic impairment compared with matched control subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe hepatic impairment or matched control
* BMI between 18.0 and 40.0 kg/m2

Exclusion Criteria:

* Evidence of acute deterioration of hepatic function within 8 weeks
* ALT or AST ≥ 5 times upper limit of normal for moderates; ALT or AST ≥ 8 times upper limit of normal for severes
* Total bilirubin > 5 mg/dl for moderates; no upper limit for severes
* Hemoglobin < 10g/dl for moderates; Hemoglobin < 9g/dl for severes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
PK Assessment | 7 days
  PK Assessment in moderate and severe hepatic impairment and matched controls.PK Assessments include plasma parameters maximum observed concentration (Cmax), time to occurrence of Cmax, area under the plasma concentration-time curve from Hour 0 to the last measurable concentration(AUC0-t), area under the plasma concentration-time curve from Hour 0 extrapolated to infinity (AUC0-∞)and systemic clearance.

SECONDARY OUTCOMES:
Safety | 7 days
  Safety Assessments evaluated through adverse events, laboratory evaluations (hematology and chemistry), vital signs, ECGs, and physical examinations, in moderate and severe hepatic impairment and matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (2):
- United States (2):
  - Trius Investigator Site 001, Orlando, Florida
  - Trius Investigator Site 002, Minneapolis, Minnesota

REFERENCES:
- [Derived] Flanagan S, Minassian SL, Morris D, Ponnuraj R, Marbury TC, Alcorn HW, Fang E, Prokocimer P. Pharmacokinetics of tedizolid in subjects with renal or hepatic impairment. Antimicrob Agents Chemother. 2014 Nov;58(11):6471-6. doi: 10.1128/AAC.03431-14. Epub 2014 Aug 18. PMID 25136024